CLINICAL TRIAL: NCT00209729
Title: Phase I/II Study of Oral S-1 Plus Docetaxel in Elderly Patients With Advanced Gastric Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Registration is less
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Responsible Party: Yoshito Komatsu / A vice-director, Associate Prof., Hokkaido University Hospital Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0502; DS-Elderly
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Gastric Cancer
Keywords: Docetaxel; S-1; Elderly Patients; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; titanium silicide; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Docetaxel plus S-1
  Interventions: Drug: Taxotere; Drug: TS-1

INTERVENTIONS:
Drug: Taxotere — X mg/m2, IV (in the vein) on day 1 and 15 of each 28 day cycle.
  Other Names: Docetaxel
Drug: TS-1 — Day 1-14, P.O. everyday
  Other Names: S-1

SUMMARY:
To assess the usefulness of Docetaxel plus S-1 combination chemotherapy based on the antitumor effect and survival period by performing a phase I/II study of this combination in Elderly patients with inoperable or with postoperative gastric cancer.

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase I/II clinical trial is conducted on Elderly patients with histological stage IV gastric cancer given Docetaxel plus S-1. The usefulness of this regimens as 1st line therapy for gastric cancer was evaluated by the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of gastric adenocarcinoma.
2. Measurable or assessable lesions(Except for Phase I).
3. Age: 76 ~ 80 years.
4. Performance Status (ECOG): 0 ~ 2.
5. No prior chemotherapy or only one regimen of previous chemotherapy (with a washout period >4 weeks after the final day of the previous therapy). Adjuvant chemotherapy is not defined as previous therapy.
6. No history of treatment with Docetaxel or S-1.
7. No history of radiotherapy to the abdomen.
8. Oral intake of S-1 is possible.
9. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and 12,000/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5 times the upper limit of normal (excluding liver metastasis). T-Bil 2.0mg/dl. Creatinine <1.5 mg/dl (but if it is 1.0 ~ 1.5 mg/dl, the dose of S-1 can be decreased according to the dose reduction criteria to allow registration in the trial). Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).
10. Predicted survival for >3 months.
11. Able to give written informed consent.

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Diarrhea (watery stools).
6. Uncontrolled ischemic heart disease.
7. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
8. Active multiple cancer.
9. Severe mental disorder.
10. Pregnancy, possible pregnancy, or breast-feeding.
11. Flucytosine treatment.
12. Judged to be ineligible for this protocol by the attending physician.

Ages: 76 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Determine the DLT(Dose Limiting Toxicity) and MTD(Maximum Tolerated Dose) in Phase I setting. Determine the clinical response rate with Recommended dose in Phase II setting. | 1-year

SECONDARY OUTCOMES:
Determine the clinical response rate of patients in Phase I setting. | 1-year
Determine the OS(Overall Survival) and DFS(Disease Free Survival). | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital (Hokkaido University Graduate School of Medicine), Sapporo, Hokkaido, Japan